CLINICAL TRIAL: NCT02501928
Title: LONG-TERM EXTENSION STUDY TO EVALUATE THE SAFETY OF FESOTERODINE IN JAPANESE PEDIATRIC SUBJECTS WITH SYMPTOMS OF DETRUSOR OVERACTIVITY ASSOCIATED WITH A NEUROLOGICAL CONDITION (NEUROGENIC DETRUSOR OVERACTIVITY) WHO HAVE COMPLETED 24 WEEKS TREATMENT IN STUDY A0221047
Brief Title: Open-label Long-term Extension Study of Fesoterodine in Japanese Subjects With Neurogenic Detrusor Overactivity.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A0221109
Record Dates: First submitted 2015-06-01; First posted 2015-07-17 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Urinary Bladder, Neurogenic
Keywords: neurogenic detrusor overactivity; fesoterodine; Japan
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fesoterodine PR 4 mg (Experimental): Fesoterodine PR 4 mg for 28 or 40 weeks in open-label treatment period
  Interventions: Drug: Fesoterodine PR 4 mg
- Fesoterodine PR 8 mg (Experimental): Fesoterodine PR 8 mg for 28 or 40 weeks in open-label treatment period
  Interventions: Drug: Fesoterodine PR 8 mg
- Fesoterodine BIC 2 mg (Experimental): Fesoterodine BIC 2 mg for 28 weeks in open-label treatment period
  Interventions: Drug: Fesoterodine BIC 2 mg
- Fesoterodine BIC 4 mg (Experimental): Fesoterodine BIC 4 mg for 28 weeks in open-label treatment period
  Interventions: Drug: Fesoterodine BIC 4 mg

INTERVENTIONS:
Drug: Fesoterodine PR 4 mg — Fesoterodine 4 mg tablet once daily for 28 or 40 weeks
  Arms: Fesoterodine PR 4 mg
Drug: Fesoterodine PR 8 mg — Fesoterodine PR 8 mg tablet once daily for 28 or 40 weeks
  Arms: Fesoterodine PR 8 mg
Drug: Fesoterodine BIC 2 mg — Fesoterodine BIC 2 mg tablet once daily for 28 weeks
  Arms: Fesoterodine BIC 2 mg
Drug: Fesoterodine BIC 4 mg — Fesoterodine BIC 4 mg tablet once daily for 28 weeks
  Arms: Fesoterodine BIC 4 mg

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of fesoterodine following once daily long-term treatment in Japanese pediatric neurogenic detrusor overactivity (NDO) subjects.

DETAILED DESCRIPTION:
This is a Phase 3, multi-center, open-label long-term extension study in Japanese NDO subjects who participated and completed in the precedent Study A0221047 which is a 24 weeks, randomized, open label study, to investigate the safety and tolerability of fesoterodine.

This study consists of a 28-week open-label treatment period followed by a 4-week follow-up. In addition, subjects in the oxybutynin arm of the precedent Study A0221047 will continue the fesoterodine treatment until Week 40 visit in this study, in order to obtain fesoterodine 1 year treatment data.

ELIGIBILITY:
Inclusion Criteria:

•Subjects who completed 24 week treatment and all visit procedures in the precedent Study A0221047

Exclusion Criteria:

* Subjects who had major protocol violation (as determined by the Sponsor) in Study A0221047
* Concomitant medications which may increase the risk to subjects or confound study results
* Other medical conditions which may increase the risk to subjects or confound study results

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- Japan (7):
  - Aichi Children's Health and Medical Center, Ōbu, Aichi-ken
  - Chiba Children's Hospital, Midori-ku Chiba-shi, Chiba
  - Fukuoka Children's Hospital, Fukuoka, Fukuoka
  - Kanagawa Children's Medical Center, Yokohama, Kanagawa
  - Osaka Women's and Children's Hospital, Izumi-shi, Osaka
  - Shizuoka Children's Hospital, Aoi-ku Shizuoka-shi, Shizuoka
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221109&StudyName=Long-term%20Extension%20Study%20To%20Evaluate%20The%20Safety%20Of%20Fesoterodine%20In%20Japanese%20Pediatric%20Subjects%20With%20Symptoms%20Of%20Detrusor%20Overactivity%20Associated%20With%20A%20Neurological%20Condition%20%28neurogenic%20Detrusor%20Overactivity%29%20Who%20Have%20Completed%2024%20Weeks%20Treatment%20In%20Study%20A0221047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This (A0221109) was a long term extension (LTE) study only among Japanese participants who participated and completed the precedent study A0221047 (NCT01557244). Per plan, efficacy outcome measures and treatment-emergent adverse events were reported using merged data of studies A0221047 and A0221109.
Pre-assignment Details: A0221047 had 2 cohorts. Cohort 1 had an active comparator phase and Cohort 2 had an efficacy phase followed by a safety extension phase for each cohort. Japanese participants from both cohorts, if consented continued in this LTE study and received the same treatment as in A0221047, per investigator judgment on safety and tolerance of participants.
Groups:
- Fesoterodine 4 Milligram (mg) Tablet: In precedent study A0221047, participants of cohort 1, with body weight greater than (>) 25 kilogram (kg), received fesoterodine 4 mg prolonged release (PR) tablet once daily for 24 weeks (12 weeks in each active comparator and safety extension phase). Only Japanese participants, who consented to continue in this LTE study, were to receive fesoterodine 4 mg PR tablet orally once daily for another 28 weeks in this LTE study.
- Fesoterodine 8 mg Tablet: In precedent study A0221047, participants of cohort 1, with body weight >25 kg, received fesoterodine 4 mg PR tablet once daily for 1 week and if well tolerated then fesoterodine 8 mg PR tablet once daily for 11 weeks in active comparator phase and 12 weeks in safety extension phase. Only Japanese participants, who consented to continue in this LTE study, were to receive fesoterodine 8 mg PR tablet orally once daily for another 28 weeks in this LTE study.
- Oxybutynin Then Fesoterodine 4 mg Tablet: In precedent study A0221047, participants of cohort 1, with body weight >25 kg, received oxybutynin tablet at daily dose per pediatric labelling in active comparator phase for 12 weeks and then fesoterodine 4 mg PR tablet in safety extension phase once daily for 12 weeks. Only Japanese participants, who consented to continue in this LTE study, were to receive fesoterodine 4 mg PR tablet orally once daily for another 40 weeks in this LTE study.
- Oxybutynin Then Fesoterodine 8 mg Tablet: In precedent study A0221047, participants of cohort 1, with body weight >25 kg, received oxybutynin tablet at daily dose per pediatric labelling in active comparator phase for 12 weeks and then fesoterodine 4 mg PR tablet once daily for 1 week and if tolerated well received 8 mg PR tablet once daily for 11 weeks in safety extension phase. Only Japanese participants, who consented to continue in this LTE study, were to receive fesoterodine 8 mg PR tablet orally once daily for another 40 weeks in this LTE study.
- Fesoterodine 2 mg Capsule: In precedent study A0220147, participants of cohort 2, with body weight less than or equal to (<=) 25 kg, received fesoterodine 2 mg beads-in-capsule (BIC) capsules orally once daily for 24 weeks (12 weeks in each efficacy and safety extension phase). Only Japanese participants, who consented to continue in this LTE study, were to receive fesoterodine 2 mg BIC capsules orally once daily for another 28 weeks in this LTE study.
- Fesoterodine 4 mg Capsule: In precedent study A0221047, participants of cohort 2, with body weight <=25 kg, received fesoterodine 2 mg BIC capsules orally once daily for 1 week and if well tolerated then fesoterodine 4 mg BIC capsules orally once daily for 11 weeks in efficacy phase and 12 weeks in safety extension phase. Only Japanese participants, who consented to continue in this LTE study, were to receive fesoterodine 4 mg BIC capsules orally once daily for another 28 weeks in this LTE study.
Period: Overall Study
Arm/Group | Fesoterodine 4 Milligram (mg) Tablet | Fesoterodine 8 mg Tablet | Oxybutynin Then Fesoterodine 4 mg Tablet | Oxybutynin Then Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Started | 0 (No participant was assigned to this arm, in this LTE study.) | 2 | 0 (No participant was assigned to this arm, in this LTE study.) | 0 (No participant was assigned to this arm, in this LTE study.) | 7 | 3
Completed | 0 | 2 | 0 | 0 | 6 | 3
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal By Parent/Guardian | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics included only those reporting arms in which at least 1 participant was assigned. Analysis population included all enrolled participants who received at least 1 dose of study medication in this LTE study.
Groups:
- Fesoterodine 8 mg Tablet: Japanese participants of cohort 1, with body weight >25 kg, who received fesoterodine 4 mg PR tablet once daily for 1 week and if well tolerated then fesoterodine 8 mg PR tablet once daily for 11 weeks in active comparator phase and for 12 weeks in safety extension phase in precedent study A0221047 and who continued to receive fesoterodine 8 mg PR tablet orally once daily for another 28 weeks in this LTE study.
- Fesoterodine 2 mg Capsule: Japanese participants of cohort 2, with body weight <=25 kg, received fesoterodine 2 mg BIC capsules orally once daily for 24 weeks (12 weeks in each efficacy and safety extension phase) in precedent study A0221047 and who continued to receive fesoterodine 2 mg BIC capsules orally once daily for another 28 weeks in this LTE study.
- Fesoterodine 4 mg Capsule: Japanese participants of cohort 2, with body weight <=25 kg, received fesoterodine 2 mg BIC capsules orally once daily for 1 week and if well tolerated then fesoterodine 4 mg BIC capsules orally once daily for 11 weeks in efficacy phase and 12 weeks in safety extension phase in precedent study A0221047 and who continued to receive fesoterodine 4 mg BIC capsules orally once daily for another 28 weeks in this LTE study.
- Total: Total of all reporting groups
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total
Number analyzed (Participants) | 2 | 7 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.50 (0.71) | 7.86 (1.68) | 7.33 (0.58) | 8.67 (2.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 3
  Male | 0 | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 7 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 7 | 3 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs): Merged Data of Studies A0221047 and A0221109
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. A treatment emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non-serious adverse events. TEAEs were summarized for each cohort (Cohort 1 and Cohort 2, irrespective of treatment received), each treatment group and the total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: Up to a maximum of 56 weeks (24 weeks of treatment in A0221047 and 32 weeks [28 weeks treatment + 4 weeks follow up post last dose] in A0221109)
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study medication in study A0221109.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Participants of cohort 1 with body weight >25 kg, who received fesoterodine 4 mg or 8 mg PR tablet orally once daily for 24 weeks (active comparator and safety extension phase) in precedent study A0221047 and then continued the same dose and dosage form of fesoterodine for 28 weeks in this LTE study.
- Cohort 2: Participants of cohort 2 with body weight <=25 kg, who received either fesoterodine 2 mg or 4 mg capsule orally once daily for 24 weeks (efficacy and safety phase) in precedent study A0221047 and then continued the same dose and dosage form of fesoterodine for 28 weeks in this LTE study.
- Fesoterodine 8 mg Tablet: Participants of cohort 1, with body weight >25 kg, who received fesoterodine 4 mg PR tablet for 1 week and if tolerated well then fesoterodine 8 mg PR tablet once daily for 11 weeks in active comparator and 12 weeks in safety extension phase in precedent study A0221047 and who continued to receive fesoterodine 8 mg PR tablet orally once daily for another 28 weeks in this LTE study.
- Fesoterodine 2 mg Capsule: Participants of cohort 2, with body weight <=25 kg, received fesoterodine 2 mg BIC capsules orally once daily for 24 weeks (12 weeks in each efficacy and safety extension phase) in precedent study and who continued to receive fesoterodine 2 mg BIC capsules orally once daily for another 28 weeks in this LTE study.
- Fesoterodine 4 mg Capsule: Participants of cohort 2, with body weight <=25 kg, received fesoterodine 2 mg BIC capsules orally once daily for 1 week and if well tolerated then fesoterodine 4 mg BIC capsules orally once daily for 11 weeks in efficacy phase and 12 weeks in safety extension phase in precedent study A0221047 and who continued to receive fesoterodine 4 mg BIC capsules orally once daily for another 28 weeks in this LTE study.
- Total of Treatment Groups: Total participants who received fesoterodine 8 mg PR tablet, fesoterodine 2 mg and 4 mg BIC capsules in precedent study A0221047 and continued to receive the same treatment respectively, in this LTE study.
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
Participants
  Participants with AEs | 2 | 9 | 2 | 6 | 3 | 11
  Participants with SAEs | 0 | 1 | 0 | 1 | 0 | 1

2. Primary Outcome: Change From Baseline in Visual Acuity at Week 12: Study A0221109
Description: Visual acuity (VA) was assessed for each eye using the Snellen method, where logarithm of minimum angle of resolution (logMAR) units were derived from the Snellen ratios. Participants had to read letters from the chart at a distance of 20 feet/6 meter or 4 meter. VA (Snellen ratio) = distance between the chart and participant, divided by distance at which participant was able to see/read chart without impairment; expressed as decimal. logMAR = log10 (1/decimal VA). In this outcome measure, data have been reported for right and left eye separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
LogMAR
  Right Eye: Baseline | 0.27 (0.376) | 0.04 (0.137) | 0.28 (0.334)
  Right Eye: Change at Week 12 | 0.14 (0.204) | -0.03 (0.083) | 0.04 (0.067)
  Left Eye: Baseline | 0.45 (0.350) | 0.04 (0.183) | 0.63 (0.663)
  Left Eye: Change at Week 12 | 0.03 (0.126) | 0.03 (0.116) | 0.07 (0.122)

3. Primary Outcome: Change From Baseline in Visual Acuity at Week 28: Study A0221109
Description: VA was assessed for each eye using the Snellen method, where logMAR units were derived from the Snellen ratios. Participants had to read letters from the chart at a distance of 20 feet/6 meter or 4 meter. VA (Snellen ratio) = distance between the chart and participant, divided by distance at which participant was able to see/read chart without impairment; expressed as decimal. logMAR = log10 (1/decimal VA). In this outcome measure, data have been reported for right and left eye separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 28
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study medication in study A0221109. Here, 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 6 | 3
LogMAR
  Right Eye | 0.00 (0.000) | 0.03 (0.118) | 0.02 (0.142)
  Left Eye | 0.31 (0.681) | 0.05 (0.057) | 0.16 (0.208)

4. Primary Outcome: Change From Baseline in Visual Acuity at Final Visit: Study A0221109
Description: as for outcome 3
Time Frame: A0221109: Baseline, Final visit (Week 28 for participants who completed the study or in case of early withdrawal the last assessment before Week 28 was considered to be the final visit)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
LogMAR
  Right Eye | 0.00 (0.000) | 0.02 (0.108) | 0.02 (0.142)
  Left Eye | 0.31 (0.681) | 0.04 (0.055) | 0.16 (0.208)

5. Primary Outcome: Change From Baseline in Visual Accommodation at Week 12: Study A0221109
Description: The visual accommodation was the minimum focusing distance for each eye at which vision became blurred - the mean of triplicate measurements. The participants focused on a single letter of the 20/40 line of an eye chart and chart was moved slowly towards the participant until letter was blurred. At this point, the distance from eye to letter was measured for each eye. In this outcome measure data have been reported for right and left eye separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study medication in study A0221109. Here, 'Number Analyzed' = participants evaluable for this outcome measure for specified rows.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
centimeter
  Right Eye: Baseline | 9.33 (8.014) | 8.62 (10.938) | 5.56 (4.857)
  Right Eye: Change at Week 12 | 2.50 (2.593) | 5.86 (13.287) | 6.67 (10.990)
  Left Eye: Baseline: number analyzed (Participants) | 2 | 7 | 2
  Left Eye: Baseline | 14.00 (13.199) | 9.86 (13.685) | 4.83 (6.835)
  Left Eye: Change at Week 12: number analyzed (Participants) | 2 | 7 | 2
  Left Eye: Change at Week 12 | -1.83 (2.593) | 3.24 (13.662) | 16.17 (23.806)

6. Primary Outcome: Change From Baseline in Visual Accommodation at Week 28: Study A0221109
Description: as for outcome 5
Time Frame: A0221109: Baseline, Week 28
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study medication in study A0221109. Here, 'Overall Number of Participants Analyzed' = participants evaluable for this outcome measure. Here, 'Number Analyzed' = participants evaluable for this outcome measure for specified rows.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 6 | 3
centimeter
  Right Eye | 5.17 (7.307) | 0.78 (2.639) | -0.11 (1.836)
  Left Eye: number analyzed (Participants) | 2 | 6 | 2
  Left Eye | 3.17 (5.421) | -0.39 (3.803) | 0.50 (0.707)

7. Primary Outcome: Change From Baseline in Visual Accommodation at Final Visit: Study A0221109
Description: as for outcome 5
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
centimeter
  Right Eye | 5.17 (7.307) | 4.38 (9.833) | -0.11 (1.836)
  Left Eye: number analyzed (Participants) | 2 | 7 | 2
  Left Eye | 3.17 (5.421) | 2.86 (9.263) | 0.50 (0.707)

8. Primary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) T Score (Derived Score) at Week 12: Study A0221109
Description: CBCL: assessed child's behavioral and emotional problems. Parent/caregiver of child answered 120 items, each on scale: 0=not true, 1=somewhat/sometimes true, 2=very/often true. 103 items were categorized in 8 domains: aggressive behavior, anxious/depressed, attention problems, rule-breaking behavior, social problems, somatic complaints, thought problems, withdrawn. Summary scores: Internalizing problems =anxious/depressed+withdrawn+somatic complaints; Externalizing problems =rule-breaking+aggressive behavior. Total problems =8 domains+other 17 items. Raw scores for each domain, summary and total problems =sum of scores of related items. Using ADM tool raw scores transformed/derived into standard T-scores, range: each domain=50-100, internalizing problems=34-100, externalizing problems=33-100, total problems=24-100. Lower T-score (8 domain,2 summary,total problems)=better outcomes. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
units on a scale
  Aggressive behavior: Baseline | 50.0 (0.00) | 52.6 (3.82) | 50.7 (1.15)
  Aggressive behavior: Change at Week 12 | 0.0 (0.00) | -0.1 (3.53) | 0.0 (0.00)
  Anxious/depressed: Baseline | 50.0 (0.00) | 52.1 (3.34) | 50.7 (0.58)
  Anxious/depressed: Change at Week 12 | 0.0 (0.00) | 0.7 (4.11) | -0.7 (0.58)
  Attention problems: Baseline | 50.0 (0.00) | 53.6 (3.55) | 53.3 (4.93)
  Attention problems: Change at week 12 | 0.0 (0.00) | -1.1 (2.34) | 0.0 (0.00)
  Rule-breaking behavior: Baseline | 50.5 (0.71) | 52.4 (3.60) | 53.3 (5.77)
  Rule-breaking behavior: Change at Week 12 | 0.0 (0.00) | -0.3 (4.11) | 0.0 (0.00)
  Social problems: Baseline | 50.0 (0.00) | 52.4 (2.70) | 54.3 (6.66)
  Social problems: Change at Week 12 | 0.0 (0.00) | 0.0 (3.65) | 0.7 (1.15)
  Somatic complaints: Baseline | 51.5 (2.12) | 53.4 (5.35) | 55.7 (4.62)
  Somatic complaints: Change at Week 12 | 1.5 (2.12) | 0.9 (1.46) | -2.3 (2.08)
  Thought problems: Baseline | 50.0 (0.00) | 50.9 (1.46) | 53.0 (4.36)
  Thought problems: Change at Week 12 | 0.0 (0.00) | 0.3 (1.70) | 0.0 (0.00)
  Withdrawn: Baseline | 50.0 (0.00) | 53.4 (4.86) | 52.7 (4.62)
  Withdrawn: Change at Week 12 | 0.0 (0.00) | -1.7 (4.54) | 0.0 (0.00)
  Externalizing problems: Baseline | 37.0 (4.24) | 47.6 (8.79) | 44.0 (10.00)
  Externalizing problems: Change at Week 12 | 0.0 (0.00) | -0.3 (6.07) | 0.0 (0.00)
  Internalizing problems: Baseline | 36.0 (4.24) | 49.0 (3.79) | 47.7 (7.51)
  Internalizing problems: Change at Week 12 | 3.0 (4.24) | 0.4 (5.00) | -4.0 (2.00)
  Total problems: Baseline | 30.5 (2.12) | 49.1 (3.67) | 46.7 (11.59)
  Total problems: Change at Week 12 | 3.0 (4.24) | -1.1 (2.12) | 0.3 (1.53)

9. Primary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) T Score (Derived Score) at Week 28: Study A0221109
Description: as for outcome 8
Time Frame: A0221109: Baseline, Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 6 | 3
units on a scale
  Aggressive behavior | 0.0 (0.00) | -2.2 (3.76) | -0.3 (0.58)
  Anxious/depressed | 0.0 (0.00) | -0.7 (4.13) | 0.3 (1.53)
  Attention problems | 0.0 (0.00) | -1.0 (2.45) | 0.0 (0.00)
  Rule-breaking behavior | -0.5 (0.71) | -1.0 (2.97) | 1.3 (2.31)
  Social problems | 0.0 (0.00) | 0.3 (1.63) | 1.0 (1.73)
  Somatic complaints | 0.0 (0.00) | 1.2 (1.83) | -2.3 (2.08)
  Thought problems | 0.0 (0.00) | -0.2 (0.41) | -0.3 (0.58)
  Withdrawn | 0.0 (0.00) | -2.0 (7.04) | 0.0 (0.00)
  Externalizing problems | -3.0 (4.24) | -3.5 (5.92) | 0.0 (0.00)
  Internalizing problems | 0.0 (0.00) | -2.5 (6.83) | -2.7 (3.06)
  Total problems | -2.5 (3.54) | -1.7 (2.94) | 1.0 (1.00)

10. Primary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) T Score (Derived Score) at Final Visit: Study A0221109
Description: as for outcome 8
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
units on a scale
  Aggressive behavior | 0.0 (0.00) | -1.9 (3.53) | -0.3 (0.58)
  Anxious/depressed | 0.0 (0.00) | -0.6 (3.78) | 0.3 (1.53)
  Attention problems | 0.0 (0.00) | -0.9 (2.27) | 0.0 (0.00)
  Rule-breaking behavior | -0.5 (0.71) | -0.9 (2.73) | 1.3 (2.31)
  Social problems | 0.0 (0.00) | 0.3 (1.50) | 1.0 (1.73)
  Somatic complaints | 0.0 (0.00) | 1.0 (1.73) | -2.3 (2.08)
  Thought problems | 0.0 (0.00) | -0.1 (0.38) | -0.3 (0.58)
  Withdrawn | 0.0 (0.00) | -1.7 (6.47) | 0.0 (0.00)
  Externalizing problems | -3.0 (4.24) | -3.0 (5.57) | 0.0 (0.00)
  Internalizing problems | 0.0 (0.00) | -2.1 (6.31) | -2.7 (3.06)
  Total problems | -2.5 (3.54) | -1.4 (2.76) | 1.0 (1.00)

11. Primary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) Total Score (Raw Score) at Week 12: Study A0221109
Description: CBCL:assessed child's behavioral and emotional problems. Parent/caregiver of child answered 120 items, each on scale:0=not true, 1=somewhat/sometimes true, 2=very/often true. 103 items were classified in 8 domains: aggressive behavior, total score range (TSR) =0-36; anxious/depressed,TSR=0-26; attention problems,TSR=0-20; rule-breaking behavior, TSR=0-34; social problems, TSR=0-22; somatic complaints, TSR=0-22; thought problems, TSR=0-30; withdrawn, TSR=0-16. Summary scores: externalizing problems combined rule-breaking and aggressive behavior,TSR=0-70; internalizing problems combined anxious/depressed, withdrawn and somatic complaints, TSR=0-64. Total problems combined 8 domains and 17 remaining items,TSR=0-240. TSR for each domain, summary and total problems was sum of scores of related items respectively. Lower scores for each domain, summary, total problems = better outcomes.Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
units on a scale
  Aggressive behavior: Baseline | 0.0 (0.00) | 3.4 (3.05) | 2.0 (2.00)
  Aggressive behavior: Change at Week 12 | 0.0 (0.00) | -0.1 (2.97) | 0.0 (0.00)
  Anxious/depressed: Baseline | 0.0 (0.00) | 1.9 (1.57) | 1.3 (1.15)
  Anxious/depressed: Change at Week 12 | 0.0 (0.00) | 0.3 (1.60) | -0.7 (0.58)
  Attention problems: Baseline | 0.0 (0.00) | 3.6 (2.64) | 3.0 (3.46)
  Attention problems: Change at week 12 | 0.0 (0.00) | -0.6 (1.27) | 0.0 (0.00)
  Rule-breaking behavior: Baseline | 0.5 (0.71) | 1.3 (1.50) | 1.3 (2.31)
  Rule-breaking behavior: Change at Week 12 | 0.0 (0.00) | -0.1 (1.21) | 0.0 (0.00)
  Social problems: Baseline | 0.0 (0.00) | 1.6 (1.27) | 2.3 (3.21)
  Social problems: Change at Week 12 | 0.0 (0.00) | 0.0 (1.63) | 0.3 (0.58)
  Somatic complaints: Baseline | 0.5 (0.71) | 1.0 (1.53) | 1.7 (1.15)
  Somatic complaints: Change at Week 12 | 0.5 (0.71) | 0.3 (0.49) | -0.7 (0.58)
  Thought problems: Baseline | 0.0 (0.00) | 0.6 (0.79) | 1.3 (1.53)
  Thought problems: Change at Week 12 | 0.0 (0.00) | -0.1 (0.69) | 0.0 (0.00)
  Withdrawn: Baseline | 0.0 (0.00) | 0.9 (1.21) | 0.7 (1.15)
  Withdrawn: Change at Week 12 | 0.0 (0.00) | -0.4 (1.13) | 0.0 (0.00)
  Externalizing problems: Baseline | 0.5 (0.71) | 4.7 (4.27) | 3.3 (4.16)
  Externalizing problems: Change at Week 12 | 0.0 (0.00) | -0.3 (3.59) | 0.0 (0.00)
  Internalizing problems: Baseline | 0.5 (0.71) | 3.7 (1.38) | 3.7 (2.31)
  Internalizing problems: Change at Week 12 | 0.5 (0.71) | 0.1 (2.19) | -1.3 (0.58)
  Total problems: Baseline | 1.5 (0.71) | 19.1 (5.79) | 18.0 (17.78)
  Total problems: Change at Week 12 | 1.0 (1.41) | -1.3 (4.07) | -0.3 (1.15)

12. Primary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) Total Score (Raw Score) at Week 28: Study A0221109
Description: as for outcome 11
Time Frame: A0221109: Baseline, Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 6 | 3
units on a scale
  Aggressive behavior | 0.0 (0.00) | -1.8 (3.06) | -0.3 (0.58)
  Anxious/depressed | 0.0 (0.00) | -0.3 (1.37) | 0.0 (1.00)
  Attention problems | 0.0 (0.00) | -0.5 (1.22) | 0.0 (0.00)
  Rule-breaking behavior | -0.5 (0.71) | -0.2 (0.98) | 0.3 (0.58)
  Social problems | 0.0 (0.00) | 0.2 (0.98) | 0.3 (0.58)
  Somatic complaints | 0.0 (0.00) | 0.3 (0.52) | -0.7 (0.58)
  Thought problems | 0.0 (0.00) | -0.2 (0.41) | -0.3 (0.58)
  Withdrawn | 0.0 (0.00) | -0.5 (1.76) | 0.0 (0.00)
  Externalizing problems | -0.5 (0.71) | -2.0 (3.58) | 0.0 (0.00)
  Internalizing problems | 0.0 (0.00) | -0.5 (2.88) | -0.7 (0.58)
  Total problems | -0.5 (0.71) | -2.7 (4.63) | 0.7 (0.58)

13. Primary Outcome: Change From Baseline in Child Behavior Checklist (CBCL) Total Score (Raw Score) at Final Visit: Study A0221109
Description: as for outcome 11
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
units on a scale
  Aggressive behavior | 0.0 (0.00) | -1.6 (2.88) | -0.3 (0.58)
  Anxious/depressed | 0.0 (0.00) | -0.3 (1.25) | 0.0 (1.00)
  Attention problems | 0.0 (0.00) | -0.4 (1.13) | 0.0 (0.00)
  Rule-breaking behavior | -0.5 (0.71) | -0.1 (0.90) | 0.3 (0.58)
  Social problems | 0.0 (0.00) | 0.1 (0.90) | 0.3 (0.58)
  Somatic complaints | 0.0 (0.00) | 0.3 (0.49) | -0.7 (0.58)
  Thought problems | 0.0 (0.00) | -0.1 (0.38) | -0.3 (0.58)
  Withdrawn | 0.0 (0.00) | -0.4 (1.62) | 0.0 (0.00)
  Externalizing problems | -0.5 (0.71) | -1.7 (3.35) | 0.0 (0.00)
  Internalizing problems | 0.0 (0.00) | -0.4 (2.64) | -0.7 (0.58)
  Total problems | -0.5 (0.71) | -2.3 (4.35) | 0.7 (0.58)

14. Primary Outcome: Change From Baseline in Grooved Pegboard Test (10 Pegs Group) at Week 12- Time to Completion: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 10 grooved pegs into holes within the given time limit up to 300 seconds. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Time taken to complete the test was inversely correlated to the cognitive ability. Participants were assigned to either a 10 or 25-peg assessment based on their age. 10-peg assessment was done on participants below age of 9 years. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study medication in study A0221109. Here "Overall Number of Participants Analyzed= participants evaluable for this outcome measure. No participant in reporting arm "Fesoterodine 8 mg Tablet" was below age of 9 years.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 5 | 3
seconds
  Dominant hand: Baseline |  | 43.0 (23.44) | 39.3 (15.18)
  Dominant hand: Change at Week 12 |  | 0.8 (6.72) | -0.3 (15.28)
  Non-dominant hand: Baseline |  | 33.4 (10.74) | 52.0 (19.67)
  Non-dominant hand: Change at Week 12 |  | 8.2 (19.93) | -1.3 (9.45)

15. Primary Outcome: Change From Baseline in Grooved Pegboard Test (10 Pegs Group) at Week 28- Time to Completion: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 10 grooved pegs into holes within the given time limit (up to 300 seconds). The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Time taken to complete the test was inversely correlated to the cognitive ability. Participants were assigned to either a 10 or 25-peg assessment based on their age. 10-peg assessment was done on participants below age of 9 years. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 28
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study medication in study A0221109. Here "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure. No participant in reporting arm "Fesoterodine 8 mg Tablet" was below age of 9 years.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 4 | 3
seconds
  Dominant hand |  | 4.5 (2.38) | 3.7 (4.04)
  Non-dominant hand |  | 6.3 (7.37) | -7.7 (10.26)

16. Primary Outcome: Change From Baseline in Grooved Pegboard Test (10 Pegs Group) at Final Visit- Time to Completion: Study A0221109
Description: as for outcome 14
Time Frame: as for outcome 4
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 5 | 3
seconds
  Dominant hand |  | 0.8 (8.53) | 3.7 (4.04)
  Non-dominant hand |  | 4.4 (7.60) | -7.7 (10.26)

17. Primary Outcome: Change From Baseline in Grooved Pegboard Test (25 Pegs Group) at Week 12- Time to Completion: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 25 grooved pegs into holes within the given time limit up to 300 seconds. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Time taken to complete the test was inversely correlated to the cognitive ability. Participants were assigned to either a 10 or 25-peg assessment based on their age. 25-peg assessment was done on participants of age 9 years and above. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study medication in study A0221109. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure. No participant in the reporting arm "Fesoterodine 4 mg Capsule" was of age 9 years and above.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 2 | 0
seconds
  Dominant hand: Baseline | 59.5 (6.36) | 107.5 (75.66) |
  Dominant hand: Change at Week 12 | 0.0 (2.83) | -11.5 (13.44) |
  Non-dominant hand: Baseline | 60.5 (6.36) | 145.5 (132.23) |
  Non-dominant hand: Change at Week 12 | -0.5 (4.95) | -2.0 (9.90) |

18. Primary Outcome: Change From Baseline in Grooved Pegboard Test (25 Pegs Group) at Week 28- Time to Completion: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 25 grooved pegs into the holes within the given time limit (up to 300 seconds). The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Time taken to complete the test was inversely correlated to the cognitive ability. Participants were assigned to either a 10 or 25-peg assessment based on their age. 25-peg assessment was done on participants of age 9 years and above. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 28
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 2 | 0
seconds
  Dominant hand | 2.0 (7.07) | -14.0 (24.04) |
  Non-dominant hand | -1.0 (2.83) | -35.0 (48.08) |

19. Primary Outcome: Change From Baseline in Grooved Pegboard Test (25 Pegs Group) at Final Visit- Time to Completion: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 25 grooved pegs into the holes within the given time limit up to 300 seconds. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Time taken to complete the test was inversely correlated to the cognitive ability. Participants were assigned to either a 10 or 25-peg assessment based on their age. 25-peg assessment was done on participants of age 9 years and above. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: as for outcome 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 2 | 0
seconds
  Dominant hand | 2.08 (7.07) | -14.0 (24.04) |
  Non-dominant hand | -1.0 (2.83) | -35.0 (48.08) |

20. Primary Outcome: Change From Baseline in Grooved Pegboard Test (10 Pegs Group) at Week 12- Number of Pegs Dropped: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 10 grooved pegs into the holes within the given time limit up to 300 seconds. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Number of pegs dropped while putting in the holes were measured. Participants were assigned to either a 10 or 25-peg assessment based on their age. 10-peg assessment was done on participants below age of 9 years. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study medication in Study A0221109. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure. No participant in reporting arm "Fesoterodine 8 mg Tablet" was below age of 9 years.
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 5 | 3
pegs
  Dominant hand: Baseline |  | 0.2 (0.45) | 0.0 (0.00)
  Dominant hand: Change at Week 12 |  | 0.2 (0.45) | 0.0 (0.00)
  Non-dominant hand: Baseline |  | 0.0 (0.00) | 0.0 (0.00)
  Non-dominant hand: Change at Week 12 |  | 0.6 (1.34) | 0.0 (0.00)

21. Primary Outcome: Change From Baseline in Grooved Pegboard Test (10 Pegs Group) at Week 28- Number of Pegs Dropped: Study A0221109
Description: as for outcome 20
Time Frame: A0221109: Baseline, Week 28
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 4 | 3
pegs
  Dominant hand |  | 0.3 (0.96) | 0.0 (0.00)
  Non-dominant hand |  | 0.0 (0.00) | 0.0 (0.00)

22. Primary Outcome: Change From Baseline in Grooved Pegboard Test (10 Pegs Group) at Final Visit- Number of Pegs Dropped: Study A0221109
Description: as for outcome 20
Time Frame: as for outcome 4
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 5 | 3
pegs
  Dominant hand |  | 0.2 (0.84) | 0.0 (0.00)
  Non-dominant hand |  | 0.0 (0.00) | 0.0 (0.00)

23. Primary Outcome: Change From Baseline in Grooved Pegboard Test (25 Pegs Group) at Week 12- Number of Pegs Dropped: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 25 grooved pegs into the holes within the given time limit up to 300 seconds. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Number of pegs dropped while putting in the holes were measured. Participants were assigned to either a 10 or 25-peg assessment based on their age. 25-peg assessment was done on participants of age 9 years and above. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 2 | 0
pegs
  Dominant hand: Baseline | 0.0 (0.00) | 0.5 (0.71) |
  Dominant hand: Change at Week 12 | 0.0 (0.00) | -0.5 (0.71) |
  Non-dominant hand: Baseline | 0.0 (0.00) | 0.5 (0.71) |
  Non-dominant hand: Change at Week 12 | 0.0 (0.00) | -0.5 (0.71) |

24. Primary Outcome: Change From Baseline in Grooved Pegboard Test (25 Pegs Group) at Week 28- Number of Pegs Dropped: Study A0221109
Description: as for outcome 23
Time Frame: A0221109: Baseline, Week 28
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 2 | 0
pegs
  Dominant hand | 0.0 (0.00) | 0.0 (1.41) |
  Non-dominant hand | 0.0 (0.00) | -0.5 (0.71) |

25. Primary Outcome: Change From Baseline in Grooved Pegboard Test (25 Pegs Group) at Final Visit- Number of Pegs Dropped: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 25 grooved pegs into the holes within the given time limit up to 300 seconds. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Number of pegs dropped while putting in the holes were measured. Participants were assigned to either a 10- or 25-peg assessment based on their age. 25-peg assessment was done on participants of age 9 years and above. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: as for outcome 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 2 | 0
pegs
  Dominant hand | 0.0 (0.00) | 0.0 (1.41) |
  Non-dominant hand | 0.0 (0.00) | -0.5 (0.71) |

26. Primary Outcome: Change From Baseline in Grooved Pegboard Test (10 Pegs Group) at Week 12- Number of Pegs Placed Correctly: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 10 grooved pegs into the holes within the given time limit up to 300 seconds. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Number of pegs placed correctly in hole was measured. Participants were assigned to either a 10 or 25-peg assessment based on their age. 10-peg assessment was done on participants below age of 9 years. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 5 | 3
pegs
  Dominant hand: Baseline |  | 10.0 (0.00) | 10.0 (0.00)
  Dominant hand: Change at Week 12 |  | 0.0 (0.00) | 0.0 (0.00)
  Non-dominant hand: Baseline |  | 10.0 (0.00) | 10.0 (0.00)
  Non-dominant hand: Change at Week 12 |  | 0.0 (0.00) | 0.0 (0.00)

27. Primary Outcome: Change From Baseline in Grooved Pegboard Test (10 Pegs Group) at Week 28- Number of Pegs Placed Correctly: Study A0221109
Description: as for outcome 26
Time Frame: A0221109: Baseline, Week 28
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 4 | 3
pegs
  Dominant hand |  | 0.0 (0.00) | 0.0 (0.00)
  Non-dominant hand |  | 0.0 (0.00) | 0.0 (0.00)

28. Primary Outcome: Change From Baseline in Grooved Pegboard Test (10 Pegs Group) at Final Visit- Number of Pegs Placed Correctly: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 10 grooved pegs into the holes within the given time limit (up to 300 seconds). The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Number of pegs placed correctly in hole was measured. Participants were assigned to either a 10 or 25-peg assessment based on their age. 10-peg assessment was done on participants below age of 9 years. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: as for outcome 4
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 5 | 3
pegs
  Dominant hand |  | 0.0 (0.00) | 0.0 (0.00)
  Non-dominant hand |  | 0.0 (0.00) | 0.0 (0.00)

29. Primary Outcome: Change From Baseline in Grooved Pegboard Test (25 Pegs Group) at Week 12- Number of Pegs Placed Correctly: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 25 grooved pegs into the holes within the given time limit up to 300 seconds. The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Number of pegs placed correctly in hole was measured. Participants were assigned to either a 10 or 25-peg assessment based on their age. 25-peg assessment was done on participants of age 9 years and above. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 2 | 0
pegs
  Dominant hand: Baseline | 25.0 (0.00) | 25.0 (0.00) |
  Dominant hand: Change at Week 12 | 0.0 (0.00) | 0.0 (0.00) |
  Non-dominant hand: Baseline | 25.0 (0.00) | 25.0 (0.00) |
  Non-dominant hand: Change at Week 12 | 0.0 (0.00) | 0.0 (0.00) |

30. Primary Outcome: Change From Baseline in Grooved Pegboard Test (25 Pegs Group) at Week 28- Number of Pegs Placed Correctly: Study A0221109
Description: The grooved pegboard test was a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. Participants were asked to insert 25 grooved pegs into the holes within the given time limit (up to 300 seconds). The task needs to be completed once for each hand; firstly, using the dominant hand followed by the non-dominant hand. Number of pegs placed correctly in hole was measured. Participants were assigned to either a 10 or 25-peg assessment based on their age. 25-peg assessment was done on participants of age 9 years and above. In this outcome measure data for dominant and non-dominant hand have been reported separately. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 28
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 2 | 0
pegs
  Dominant hand | 0.0 (0.00) | 0.0 (0.00) |
  Non-dominant hand | 0.0 (0.00) | 0.0 (0.00) |

31. Primary Outcome: Change From Baseline in Grooved Pegboard Test (25 Pegs Group) at Final Visit- Number of Pegs Placed Correctly: Study A0221109
Description: as for outcome 29
Time Frame: as for outcome 4
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: pegs
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 2 | 0
pegs
  Dominant hand | 0.0 (0.00) | 0.0 (0.00) |
  Non-dominant hand | 0.0 (0.00) | 0.0 (0.00) |

32. Primary Outcome: Change From Baseline in Vital Sign (Blood Pressure) at Week 12: Study A0221109
Description: Systolic and diastolic blood pressure were evaluated for examination of vital signs. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
millimeter of mercury
  Systolic blood pressure | 6.0 (4.24) | 2.1 (9.65) | 5.0 (14.11)
  Diastolic blood pressure | 10.5 (4.95) | -0.9 (8.90) | 6.3 (15.31)

33. Primary Outcome: Change From Baseline in Vital Sign (Blood Pressure) at Week 28: Study A0221109
Description: as for outcome 32
Time Frame: A0221109: Baseline, Week 28
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study medication in study A0221109. Here, "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 6 | 3
millimeter of mercury
  Systolic blood pressure | 8.5 (16.26) | 5.7 (11.18) | 9.7 (2.52)
  Diastolic blood pressure | 12.0 (4.24) | 5.3 (9.03) | 10.7 (2.52)

34. Primary Outcome: Change From Baseline in Vital Sign (Blood Pressure) at Final Visit: Study A0221109
Description: as for outcome 32
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millimeter of mercury
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
millimeter of mercury
  Systolic blood pressure | 8.5 (16.26) | 5.1 (10.30) | 9.7 (2.52)
  Diastolic blood pressure | 12.0 (4.24) | 4.6 (8.48) | 10.7 (2.52)

35. Primary Outcome: Change From Baseline in Vital Sign (Pulse Rate) at Week 12: Study A0221109
Description: Pulse rate was evaluated for examination of vital signs. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
beats per minute | 0.0 (18.38) | 2.4 (12.53) | -8.0 (2.00)

36. Primary Outcome: Change From Baseline in Vital Sign (Pulse Rate) at Week 28: Study A0221109
Description: as for outcome 35
Time Frame: A0221109: Baseline, Week 28
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 6 | 3
beats per minute | -3.5 (6.36) | -2.7 (8.82) | -3.7 (9.61)

37. Primary Outcome: Change From Baseline in Vital Sign (Pulse Rate) at Final Visit: Study A0221109
Description: as for outcome 35
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
beats per minute | -3.5 (6.36) | -1.4 (8.70) | -3.7 (9.61)

38. Primary Outcome: Number of Participants With Adverse Event Urinary Tract Infections (UTI): Merged Data of Studies A0221047 and A0221109
Description: UTI data were summarized for each cohort, each treatment group and the total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
Participants | 0 | 1 | 0 | 1 | 0 | 1

39. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: Hematology: hemoglobin, hematocrit, erythrocytes <0.8*lower limit of normal (LLN); platelets<0.5*LLN>1.75*upper limit of normal (ULN); leukocytes <0.6*LLN>1.5*ULN; lymphocytes, neutrophils <0.8*LLN >1.2*UL; basophils, eosinophils, monocytes >1.2*ULN. Clinical chemistry: bilirubin, direct bilirubin >1.5*ULN; aspartate aminotransferase (AT), alanine AT, gamma glutamyl transferase, lactate dehydrogenase, alkaline phosphatase >3.0*ULN; protein, albumin <0.8*LLN >1.2*ULN; blood urea nitrogen, creatinine >1.3*ULN; urate >1.2*ULN, sodium<0.95*LLN>1.05*ULN; potassium, chloride, bicarbonate <0.9*LLN>1.1*ULN; glucose <0.6*LLN>1.5*ULN; creatine kinase >2.0*ULN. Urinalysis: specific gravity <1.003>1.030, pH <4.5>8, glucose, ketones, protein, hemoglobin, nitrite, leukocyte esterase >=1; erythrocytes, leukocytes >=20; epithelial cells >=6, bacteria >20, hyaline casts >1. Data for this outcome was planned to be analysed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline to 28 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 2 | 7 | 3
Participants | 2 | 6 | 2

40. Primary Outcome: Change From Baseline in Post-Void Residual (PVR) Volume at Week 12: Study A0221109
Description: Post-void residual volume was assessed by an ultrasound. PVR volume was assessed only in participants who did not perform clean intermittent catheterization or in any participants who had >1 UTI during the study. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 12
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study medication in study A0221109. All participants performed clean intermittent catheterization, hence were not eligible for post-void residual volume assessment.
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 0 | 0

41. Primary Outcome: Change From Baseline in Post-Void Residual (PVR) Volume at Week 28: Study A0221109
Description: Post-void residual volume measurement was measured by an ultrasound. PVR volume was only assessed for participants who did not perform clean intermittent catheterization or in any participants who had >1 UTI during the study. Data for this outcome measure was planned to be analyzed for each treatment group of study A0221109 only.
Time Frame: A0221109: Baseline, Week 28
Population: as for outcome 40
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 0 | 0

42. Primary Outcome: Change From Baseline in Post-Void Residual (PVR) Volume at Final Visit: Study A0221109
Description: as for outcome 41
Time Frame: as for outcome 4
Population: as for outcome 40
Arm/Group | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule
Number analyzed (Participants) | 0 | 0 | 0

43. Secondary Outcome: Change From Baseline in Maximum Cystometric Bladder Capacity at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: Maximum cystometric bladder capacity was defined as maximal tolerable cystometric capacity, until voiding or leaking begins or at a pressure of >=40 centimeter (cm) water (H2O). Maximum cystometric bladder capacity was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: Study A0221047: Baseline, Week 12; Study A0221109: Week 28, Final Visit (Week 28 for participants who completed the study or in case of early withdrawal the last assessment before Week 28 was considered to be the final visit)
Population: Full analysis set (FAS) included all participants who were enrolled and received at least one dose of study medication and had at least 1 observation in efficacy endpoint data after baseline visit in study A0221109. Here, 'Number Analyzed' = participants evaluable for this outcome measure for specified rows.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
milliliter
  Baseline | 181.0 (28.28) | 135.5 (45.21) | 181.0 (28.28) | 149.7 (38.49) | 102.3 (48.95) | 143.1 (45.37)
  Change at Week 12 | 153.0 (56.57) | 42.9 (31.01) | 153.0 (56.57) | 37.6 (28.83) | 55.3 (38.76) | 61.3 (53.98)
  Change at Week 28: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Week 28 | 121.5 (30.41) | 37.9 (53.99) | 121.5 (30.41) | 32.8 (52.42) | 48.0 (67.55) | 53.1 (59.74)
  Change at Final Visit: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Final Visit | 121.5 (30.41) | 37.9 (53.99) | 121.5 (30.41) | 32.8 (52.42) | 48.0 (67.55) | 53.1 (59.74)

44. Secondary Outcome: Change From Baseline in Detrusor Pressure at Maximum Bladder Capacity at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: Detrusor pressure (cm H2O) at maximum urinary bladder capacity was measured using urodynamic testing. Detrusor pressure was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: FAS included all participants who were enrolled and received at least one dose of study medication and had at least 1 observation in efficacy endpoint data after baseline visit in study A0221109. Here, 'Number Analyzed' = participants evaluable for this outcome measure for specified rows.
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
cm H2O
  Baseline | 29.0 (8.49) | 40.2 (31.34) | 29.0 (8.49) | 32.4 (11.57) | 58.3 (57.55) | 38.3 (28.79)
  Change at Week 12 | -5.5 (0.71) | -13.7 (24.90) | -5.5 (0.71) | -6.0 (7.85) | -31.7 (43.73) | -12.3 (22.74)
  Change at Week 28: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Week 28 | -7.0 (0.00) | -4.3 (23.93) | -7.0 (0.00) | -2.8 (2.86) | -7.3 (47.44) | -4.8 (21.43)
  Change at Final Visit: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Final Visit | -7.0 (0.00) | -4.3 (23.93) | -7.0 (0.00) | -2.8 (2.86) | -7.3 (47.44) | -4.8 (21.43)

45. Secondary Outcome: Number of Participants With Presence of Involuntary Detrusor Contraction (IDC) at Baseline and Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: Participants with presence of IDC was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: FAS included all participants who were enrolled and received at least one dose of study medication and had at least 1 observation in efficacy endpoint data after baseline visit in study A0221109.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
Participants
  Baseline | 1 | 10 | 1 | 7 | 3 | 11
  Week 12 | 0 | 7 | 0 | 4 | 3 | 7
  Week 28 | 0 | 8 | 0 | 5 | 3 | 8
  Final Visit | 0 | 8 | 0 | 5 | 3 | 8

46. Secondary Outcome: Change From Baseline in Bladder Volume at First Involuntary Detrusor Contraction (IDC) at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: Bladder volume at first IDC was measured using urodynamic testing. Bladder volume at first IDC was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: FAS included all participants who were enrolled and received at least one dose of study medication and had at least 1 observation in efficacy endpoint data after baseline visit. Overall number of participants analyzed=participants evaluable for this outcome measure. Number Analyzed=participants evaluable for this outcome measure for specified rows.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 1 | 10 | 1 | 7 | 3 | 11
milliliter
  Baseline | 175.0 | 48.8 (31.65) | 175.0 | 48.1 (36.57) | 50.3 (22.14) | 60.3 (48.47)
  Change at Week 12: number analyzed (Participants) | 0 | 7 | 0 | 4 | 3 | 7
  Change at Week 12 |  | 95.0 (53.88) |  | 113.8 (68.55) | 70.0 (4.58) | 95.0 (53.88)
  Change at Week 28: number analyzed (Participants) | 0 | 8 | 0 | 5 | 3 | 8
  Change at Week 28 |  | 50.4 (36.38) |  | 38.6 (24.46) | 70.0 (50.11) | 50.4 (36.38)
  Change at Final Visit: number analyzed (Participants) | 0 | 8 | 0 | 5 | 3 | 8
  Change at Final Visit |  | 50.4 (36.38) |  | 38.6 (24.46) | 70.0 (50.11) | 50.4 (36.38)

47. Secondary Outcome: Change From Baseline in Bladder Compliance at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: Bladder compliance was defined as change in bladder volume in milliliter (mL) divided by change in bladder pressure in cm H2O (during the same time when change in bladder volume was estimated). Bladder Compliance was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: milliliter per cm H2O
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
milliliter per cm H2O
  Baseline | 7.00 (2.828) | 6.97 (5.124) | 7.00 (2.828) | 8.16 (5.668) | 4.20 (2.307) | 6.98 (4.712)
  Change at Week 12 | 9.00 (7.071) | 20.06 (46.151) | 9.00 (7.071) | 23.34 (55.493) | 12.40 (14.855) | 18.22 (42.021)
  Change at Week 28: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Week 28 | 8.65 (6.152) | 13.22 (16.721) | 8.65 (6.152) | 13.18 (18.628) | 13.30 (15.836) | 12.39 (15.194)
  Change at Final Visit: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Final Visit | 8.65 (6.152) | 13.22 (16.721) | 8.65 (6.152) | 13.18 (18.628) | 13.30 (15.836) | 12.39 (15.194)

48. Secondary Outcome: Change From Baseline in Mean Number of Micturitions Per 24 Hours at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: The mean number of micturitions per 24 hours were calculated as the total number of micturitions divided by the total number of diary days collected at the assessment time point. Number of diary days collected at the assessment time point = number of calendar days when the diary was completed on, even if it was not a full 24 hour period. This outcome measure was only calculated for participants with >0 micturitions at Baseline. Data was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: FAS was analyzed. Here "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure. No participant in reporting arms "Cohort 1", "Fesoterodine 8 mg Tablet" and "Fesoterodine 4 mg Capsule" had >0 micturitions at baseline.
Measure: Mean (Standard Deviation); unit: micturitions per 24 hours
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 0 | 4 | 0 | 4 | 0 | 4
micturitions per 24 hours
  Baseline |  | 4.58 (4.541) |  | 4.58 (4.541) |  | 4.58 (4.541)
  Change at Week 12 |  | -1.50 (1.036) |  | -1.50 (1.036) |  | -1.50 (1.036)
  Change at Week 28 |  | -1.08 (0.631) |  | -1.08 (0.631) |  | -1.08 (0.631)
  Change at Final Visit |  | -1.08 (0.631) |  | -1.08 (0.631) |  | -1.08 (0.631)

49. Secondary Outcome: Change From Baseline in Mean Number of Catheterizations Per 24 Hours at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: The mean number of catheterizations per 24 hours were calculated as the total number of catheterizations divided by the total number of diary days collected at the assessment time point. Number of diary days collected at the assessment time point = number of calendar days when the diary was completed, even if it was not a full 24 hour period. This outcome measure was only calculated for participants with >0 catheterizations at Baseline. Data was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: catheterizations per 24 hours
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
catheterizations per 24 hours
  Baseline | 5.33 (0.943) | 4.47 (1.390) | 5.33 (0.943) | 4.24 (1.641) | 5.00 (0.000) | 4.61 (1.332)
  Change at Week 12 | 0.00 (0.471) | 0.05 (0.357) | 0.00 (0.471) | 0.03 (0.420) | 0.11 (0.192) | 0.04 (0.353)
  Change at Week 28: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Week 28 | 0.33 (0.000) | -0.09 (0.278) | 0.33 (0.000) | -0.19 (0.267) | 0.11 (0.192) | -0.02 (0.302)
  Change at Final Visit | 0.33 (0.000) | -0.12 (0.273) | 0.33 (0.000) | -0.21 (0.249) | 0.11 (0.192) | -0.04 (0.303)

50. Secondary Outcome: Change From Baseline in Mean Number of Micturitions or Catheterizations Combined Per 24 Hours at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: The mean number of micturitions and catheterizations combined per 24 hours were calculated as the total number of micturitions and catheterizations combined divided by the total number of diary days collected at the assessment point. Number of diary days collected at the assessment time point = number of calendar days when the diary was completed, even if it was not a full 24 hour (hr) period. This outcome measure was only calculated for participants with >0 micturitions or catheterizations at Baseline. Data was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: micturitions or catheterizations/24 hr
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
micturitions or catheterizations/24 hr
  Baseline | 5.33 (0.943) | 6.30 (2.808) | 5.33 (0.943) | 6.86 (3.259) | 5.00 (0.000) | 6.14 (2.584)
  Change at Week 12 | 0.00 (0.471) | -0.55 (1.131) | 0.00 (0.471) | -0.83 (1.264) | 0.11 (0.192) | -0.46 (1.055)
  Change at Week 28: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Week 28 | 0.33 (0.000) | -0.57 (0.741) | 0.33 (0.000) | -0.92 (0.665) | 0.11 (0.192) | -0.41 (0.758)
  Change at Final Visit | 0.33 (0.000) | -0.55 (0.703) | 0.33 (0.000) | -0.83 (0.645) | 0.11 (0.192) | -0.40 (0.723)

51. Secondary Outcome: Change From Baseline in Mean Number of Incontinence Episodes Per 24 Hours at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: The mean number of incontinence episodes per 24 hours were calculated as the total number of incontinence episodes divided by the total number of diary days collected at the assessment time point. Number of diary days collected at the assessment time point = number of calendar days when the diary was completed, even if it was not a full 24 hour period. This outcome measure was only calculated for participants with >0 incontinence episodes at Baseline. Data was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: incontinence episodes per 24 hours
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
incontinence episodes per 24 hours
  Baseline | 1.17 (0.236) | 3.60 (2.298) | 1.17 (0.236) | 3.48 (2.768) | 3.89 (0.770) | 3.19 (2.285)
  Change at Week 12 | 0.50 (0.236) | -0.18 (1.726) | 0.50 (0.236) | -0.26 (2.074) | 0.00 (0.667) | -0.07 (1.586)
  Change at Week 28: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Week 28 | 1.83 (0.707) | -0.31 (1.501) | 1.83 (0.707) | -0.42 (1.577) | -0.11 (1.644) | 0.08 (1.615)
  Change at Final Visit | 1.83 (0.707) | 0.08 (1.894) | 1.83 (0.707) | 0.17 (2.110) | -0.11 (1.644) | 0.38 (1.856)

52. Secondary Outcome: Change From Baseline in Mean Number of Urgency Episodes Per 24 Hours at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: The mean number of urgency episodes per 24 hours were calculated as the total number of urgency episodes divided by the total number of diary days collected at the assessment time point. Number of diary days collected at the assessment time point = number of calendar days when the diary was completed, even if it was not a full 24 hour period. Urgency episodes were defined as urgency marked as 'yes' in the diary. This outcome measure was only calculated for sensate participants with >0 urgency episodes at Baseline. Data was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: FAS was analyzed. Here "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure. No sensate participants for reporting arms "Cohort 1" and "Fesoterodine 8 mg Tablet" had >0 urgency episodes at baseline.
Measure: Mean (Standard Deviation); unit: urgency episodes per 24 hours
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 0 | 3 | 0 | 2 | 1 | 3
urgency episodes per 24 hours
  Baseline |  | 0.61 (0.347) |  | 0.75 (0.354) | 0.33 | 0.61 (0.347)
  Change at Week 12 |  | -0.61 (0.347) |  | -0.75 (0.354) | -0.33 | -0.61 (0.347)
  Change at Week 28 |  | -0.61 (0.347) |  | -0.75 (0.354) | -0.33 | -0.61 (0.347)
  Change at Final Visit |  | -0.61 (0.347) |  | -0.75 (0.354) | -0.33 | -0.61 (0.347)

53. Secondary Outcome: Change From Baseline in Mean Volume Voided Per Micturition at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: The mean voided volume per micturition was calculated as sum of voided volume divided by the total number of micturition episodes with a recorded voided volume >0. This outcome measure included only participants who actually had the records of volume voided per micturition. Data was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: FAS was analyzed. Here "Overall Number of Participants Analyzed"= participants evaluable for this outcome measure. No participant in reporting arms "Cohort 1", "Fesoterodine 8 mg Tablet" and "Fesoterodine 4 mg Capsule" had the records of volume voided per micturition.
Measure: Mean (Standard Deviation); unit: milliliter per micturition
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 0 | 2 | 0 | 2 | 0 | 2
milliliter per micturition
  Baseline |  | 73.42 (42.309) |  | 73.42 (42.309) |  | 73.42 (42.309)
  Change at Week 12 |  | 15.77 (6.924) |  | 15.77 (6.924) |  | 15.77 (6.924)
  Change at Week 28 |  | 4.75 (14.496) |  | 4.75 (14.496) |  | 4.75 (14.496)
  Change at Final Visit |  | 4.75 (14.496) |  | 4.75 (14.496) |  | 4.75 (14.496)

54. Secondary Outcome: Change From Baseline in Mean Volume Voided Per Catheterization at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: The mean volume per catheterization was calculated as sum of voided volume divided by the total number of catheterization, with a recorded voided volume >0. This outcome measure included only participants who actually had the records of volume voided per catherization. Data was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: milliliter per catheterization
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
milliliter per catheterization
  Baseline | 198.75 (44.194) | 58.31 (40.187) | 198.75 (44.194) | 48.76 (39.230) | 80.58 (39.841) | 81.72 (66.988)
  Change at Week 12 | -0.92 (21.095) | 20.66 (21.024) | -0.92 (21.095) | 17.90 (17.038) | 27.08 (32.086) | 17.06 (21.739)
  Change at Week 28: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Week 28 | -29.42 (12.139) | 11.58 (27.064) | -29.42 (12.139) | 8.72 (33.245) | 17.28 (9.659) | 4.12 (29.591)
  Change at Final Visit: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Final Visit | -29.42 (12.139) | 11.58 (27.064) | -29.42 (12.139) | 8.72 (33.245) | 17.28 (9.659) | 4.12 (29.591)

55. Secondary Outcome: Change From Baseline in Mean Volume Voided Per Micturition or Catheterization at Week 12 of Study A0221047 and at Week 28 and Final Visit of Study A0221109
Description: The mean voided volume per micturition or catheterization was calculated as sum of voided volume divided by the total number of micturition or catheterization episodes with a recorded voided volume >0. Data was summarized for each cohort, each treatment group and total of treatment groups, using the merged data of studies A0221047 and A0221109 as planned.
Time Frame: as for outcome 43
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: mL per micturition or catheterization
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
Number analyzed (Participants) | 2 | 10 | 2 | 7 | 3 | 12
mL per micturition or catheterization
  Baseline | 198.75 (44.194) | 65.68 (34.769) | 198.75 (44.194) | 59.29 (33.550) | 80.58 (39.841) | 87.86 (62.045)
  Change at Week 12 | -0.92 (21.095) | 17.88 (17.597) | -0.92 (21.095) | 13.94 (7.801) | 27.08 (32.086) | 14.75 (18.638)
  Change at Week 28: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Week 28 | -29.42 (12.139) | 12.34 (26.812) | -29.42 (12.139) | 9.86 (33.029) | 17.28 (9.659) | 4.75 (29.583)
  Change at Final Visit: number analyzed (Participants) | 2 | 9 | 2 | 6 | 3 | 11
  Change at Final Visit | -29.42 (12.139) | 12.34 (26.812) | -29.42 (12.139) | 9.86 (33.029) | 17.28 (9.659) | 4.75 (29.583)

ADVERSE EVENTS:
Time Frame: Up to a maximum of 56 weeks (24 weeks of treatment in A0221047 and 32 weeks [28 weeks treatment + 4 weeks follow up post last dose] in A0221109)
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis population evaluated. AEs were summarized for each cohort (Cohort 1 and Cohort 2), each treatment group and the total of treatment groups , using the merged data of studies A0221047 and A0221109 as planned.
Arm/Group | Cohort 1 | Cohort 2 | Fesoterodine 8 mg Tablet | Fesoterodine 2 mg Capsule | Fesoterodine 4 mg Capsule | Total of Treatment Groups
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/10 | 0/2 | 0/7 | 0/3 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/10 | 0/2 | 1/7 | 0/3 | 1/12
Other Adverse Events (participants affected / at risk) | 2/2 | 9/10 | 2/2 | 6/7 | 3/3 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=2) | Cohort 2 (N=10) | Fesoterodine 8 mg Tablet (N=2) | Fesoterodine 2 mg Capsule (N=7) | Fesoterodine 4 mg Capsule (N=3) | Total of Treatment Groups (N=12)
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=2) | Cohort 2 (N=10) | Fesoterodine 8 mg Tablet (N=2) | Fesoterodine 2 mg Capsule (N=7) | Fesoterodine 4 mg Capsule (N=3) | Total of Treatment Groups (N=12)
Astigmatism (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1
Myopia (Eye disorders) | 0 | 2 | 0 | 0 | 2 | 2
Strabismus (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 2
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 1 | 1 | 1 | 3
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 0 | 4 | 0 | 3 | 1 | 4
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 6 | 1 | 4 | 2 | 7
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 2
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 2
Chillblains (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 1
Urodynamics measurement abnormal (Investigations) | 0 | 1 | 0 | 0 | 1 | 1
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 1
Device malfunction (Product Issues) | 0 | 1 | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 1 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
Prioritization of outcome measures was based on study team's discretion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-01-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT02501928/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT02501928/SAP_001.pdf